CLINICAL TRIAL: NCT02806778
Title: Monitoring of Cerebral Oxygenation Using Jugular Oximetry in Comatose Patients After Cardiac Arrest
Status: Completed | Type: Observational
Sponsor: University Hospital Ostrava (Other)
Responsible Party: Sponsor
Other Study IDs: FNO-KARIM-4
Record Dates: First submitted 2016-06-16; First posted 2016-06-21 (Estimated); Last update posted 2019-03-29 (Actual); Status verified 2019-03

CONDITIONS: Cerebral Hypoxic Injury; Cardiac Arrest
Keywords: cardiac arrest; jugular venous oximetry; hypoxic brain injury
MeSH Terms: conditions — Heart Arrest; Hypoxia, Brain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hypoxic brain injury: Consecutive out-of-hospital, post-cardiac arrest patients who remain comatose after successful resuscitation, admitted on ICU of University Hospital Ostrava. The patients will undergo BIS monitor-guided sedation and jugular bulb catheterisation.
  Interventions: Other: BIS Monitor-guided sedation; Other: Jugular bulb catheter

INTERVENTIONS:
Other: BIS Monitor-guided sedation — The patients enrolled in the study will undergo BIS Monitor-guided sedation. Standard BIS Monitor will be used for the procedure to monitor the depth of sedation.
Other: Jugular bulb catheter — Jugular bulb catheter will be implanted in the patients enrolled in the study.

SUMMARY:
The use of protective ventilation (to maintain normoxia and normocapnia), optimise haemodynamics, diagnose/treat seizures, therapeutic hypotermia etc is recommended for ICU management of patients who have had cardiac arrest and remain in coma after return of spontaneous circulation according to the latest International Guidelines. These actions essentially aim to limit secondary brain injury but despite all therapeutic effort, the cerebral oxygenation may remain inadequate and there is no validated method to avoid such a state in real time.

DETAILED DESCRIPTION:
The use of protective ventilation (to maintain normoxia and normocapnia), optimize hemodynamics, diagnose/treat seizures, therapeutic hypothermia etc is recommended for ICU management of patients who have had cardiac arrest and remain in a coma after the return of spontaneous circulation according to the latest International Guidelines. These actions essentially aim to limit secondary brain injury but despite all therapeutic effort, the cerebral oxygenation may remain inadequate and there is no validated method to avoid such a state in real time.

The objective of this study is to assess the relationship between jugular venous oximetry and neurological outcome of comatose patients after cardiac arrest, evaluated as per the Cerebral Performance Category scale (CPC). Further, the aim is to clarify relations between biomarkers protein S100B, neuron-specific enolase (NSE) and parameters of jugular oximetry for prognostication. An anticipated total of sixty patients will be enrolled in this non-randomised, single-group, double-blind study.

In the course of the study, the authors have decided to stop using BIS monitoring for sedation management. Reason for this decision was very limited reliability of this technique in unparalyzed patients on ICU (muscle artifacts). New aim of sedation was Richmond Agitation Sedation Scale (RASS) -4 or -5, with avoiding shivering and clinically manifested seizures.

ELIGIBILITY:
Inclusion Criteria:

* age 18 or older
* successful cardiopulmonary resuscitation
* persistent coma defined as: no eye opening to voice and inability to follow commands

Exclusion Criteria:

* pre-existing "do not resuscitate" status
* severe coexisting systemic disease with a limited life expectancy
* pregnancy
* patients who will die within 72 h of the initial cardiac arrest

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive out-of-hospital, post-cardiac arrest patients who remain comatose after successful resuscitation, admitted on ICU University Hospital Ostrava will be enrolled into the study.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2016-06; Primary Completion 2018-06 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Oxygen Saturation of Jugular Venous Bulb | 24 months
  The saturation of oxygen will be monitored after admission to ICU and every 6 hours for the total period of 72 hour after cardiac arrest
Serum S100B level | 24 months
  The serum S100B level will be monitored after admission of the patients to ICU
Serum NSE level | 24 months
  The serum NSE level will be monitored after admission of the patient to ICU and 24, 48 and 72 hour after cardiac arrest
BIS monitor guided sedation to level 40-60 | 24 months
  BIS monitor-guided sedation with the aim of achieving the level of 40-60 will be maintained for 36 hour after admission of the patients to ICU

SECONDARY OUTCOMES:
Functional status | 24 months
  Functional status defined with using cerebral performance category (CPC) classification will be assessed at time of discharge from the hospital and at 3 months after cardiac arrest

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Ostrava, Ostrava-Poruba, Moravian-Silesian Region, Czechia

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be made available. The results of the study will be published in an impact factor journal.